CLINICAL TRIAL: NCT07266350
Title: A Non-interventional Registration Study of Monotherapy or Combination Regimens Based on Camrelizumab or Famitinib for the Treatment of Cervical Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Qi Zhou (Other)
Responsible Party: Sponsor-Investigator, Qi Zhou, doctor, Chongqing University Cancer Hospital
Organization: Chongqing University Cancer Hospital (Other)
Other Study IDs: CZLL2025-042-001
Record Dates: First submitted 2025-11-16; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Cervical Cancer Metastatic; Cervical Cancer Recurrent
MeSH Terms: interventions — camrelizumab; famitinib

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Cohort 1: camrelizumab
  Interventions: Drug: Camrelizumab
- Cohort 2: famitinib
  Interventions: Drug: Famitinib
- Cohort 3: camrelizumab +famitinib
  Interventions: Drug: Camrelizumab; Drug: Famitinib
- Cohort 4: camrelizumab+others
  Interventions: Drug: Camrelizumab
- Cohort 5: famitinib+others
  Interventions: Drug: Famitinib
- Cohort 6: camrelizumab+famitinib+others
  Interventions: Drug: Camrelizumab; Drug: Famitinib

INTERVENTIONS:
Drug: Camrelizumab — 200mg IV Q3W
  Groups: Cohort 1; Cohort 3; Cohort 4; Cohort 6
Drug: Famitinib — 20mg QD PO
  Groups: Cohort 2; Cohort 3; Cohort 5; Cohort 6

SUMMARY:
This trial is a national multicenter, open-label, non-interventional study to observe and evaluate the safety and efficacy of monotherapy or combination regimens based on camrelizumab or famitinib in patients with cervical cancer.

This study included patients with cervical cancer who used monotherapy or combination regimens based on camrelizumab or famitinib. The administration regimens include but are not limited to camrelizumab monotherapy, camrelizumab in combination with mitinib, famitinib monotherapy, camrelizumab in combination with other treatment regimens selected by the investigator, camrelizumab in combination with mitinib and other treatment regimens selected by the investigator, and famitinib in combination with other treatment regimens selected by the investigator.

It is planned to include cervical cancer patients who have decided to be treated with monotherapy or combination regimens based on camrelizumab or famitinib before enrollment, with an estimated 1,300 cases.

According to the treatment plan received by the patients, after enrollment, they can be respectively placed in one of the following six cohorts:

Queue 1: Only receiving camrelizumab monotherapy

Queue 2: Only receiving famitinib monotherapy

Queue 3: Only combination therapy of camrelizumab and famitinib was received

Queue 4: Receiving camrelizumab in combination with other treatment regimens

Queue 5: Receiving famitinib in combination with other treatment regimens

Queue 6: Receiving camrelizumab and famitinib in combination with other treatment regimens

Data from the baseline period, treatment period and follow-up period were collected respectively according to the cohort category (prospective or retrospective) of the enrolled patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old;
2. Sign the informed consent form and voluntarily join this study;
3. Patients with cervical cancer diagnosed by histopathology;
4. Receive treatment with monotherapy or combination regimens based on camrelizumab or famitinib;
5. It is necessary to agree to take effective contraceptive measures and avoid egg donation from the time of signing the informed consent form until 2 months after the last administration of camrelizumab, 3 months after the last administration of famitinib, or within the contraceptive period specified in the instructions of the last administration of other study drugs (whichever is longer).

If a patient has had menstruation but has not yet reached postmenopausal status (with no menstruation for a continuous period of ≥12 months and no other causes found except menopause), and has not undergone sterilization surgery (such as hysterectomy, bilateral tubal ligation or bilateral oophorectomy), the patient is considered to have fertility.

Exclusion Criteria:

1. There is already evidence indicating that the patient is a pregnant or lactating woman.
2. Currently participating in any research involving intervention measures outside of regular clinical practice;
3. The researcher determines other circumstances that are not suitable for inclusion in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with confirmed cervical cancer
Sampling Method: Probability Sample
Enrollment: 1300 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2028-12-30 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
safety according to CTCAE v5.0 | From the first administration to 30 days after the end of the medication
  The safety of monotherapy or combination regimens based on camrelizumab or famitinib in patients with cervical cancer under real-world conditions. Per CTCAE v5.0, preferred term and grade will be documented.

SECONDARY OUTCOMES:
real world ORR | from the initiation of monotherapy or combination regimens, per 6-8 weeks
  It is defined as the sum of the proportions of patients with complete response (CR) and partial response (PR) based on investigator assessment from the initiation of monotherapy or combination regimens based on camrelizumab or famitinib to disease progression/recurrence or the start of new anti-tumor treatment.
overall survival | From date of treatment until the date of date of death from any cause, assessed up to 3 years
  It is defined as the time from the start of the first treatment to death caused by any reason.

CONTACTS AND LOCATIONS:
Overall Officials: qi zhou, Principal Investigator — Chongqing University Cancer Hospital & Chongqing Cancer Institute & Chongqing Cancer Hospital,